CLINICAL TRIAL: NCT00661791
Title: Effects of Massage Therapy and Kinesthetic Stimulation on Pre-Term Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: George Washington University (Other)
Responsible Party: Hany Z. Aly, MD, George Washington University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB120206
Record Dates: First submitted 2008-04-15; First posted 2008-04-18 (Estimated); Last update posted 2008-04-18 (Estimated); Status verified 2008-04

CONDITIONS: Prematurity
Keywords: preterm infants; massage; physical activity; weight gain; length of hospital stay; NICU
MeSH Terms: conditions — Premature Birth; Motor Activity; Weight Gain | interventions — Massage; Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- A (No Intervention): Control Group receives routine care.
- B. (Experimental): massage group, receives massage only.
  Interventions: Behavioral: Massage therapy without exercise
- C. (Experimental): Massage and Exercise group, receives both massage and exercise.
  Interventions: Behavioral: Massage therapy with exercise

INTERVENTIONS:
Behavioral: Massage therapy without exercise — Infants will receive massage twice a day; 15 minutes each.
  Arms: B.
Behavioral: Massage therapy with exercise — Infants will receive massage with exercise twice a day; 15 minutes each.
  Arms: C.

SUMMARY:
The purpose of this study was to determine whether massage with or without physical exercise impacted weight gain or length of hospital stay for premature infants.

DETAILED DESCRIPTION:
Premature infants are often cared for in a fashion that minimizes physical activity in order to reduce stress and stress-related complications. Previous studies have indicated that massage therapy may increase weight gain and enabled earlier discharge of premature infants.

In this study, premature infants were randomly assigned to one of three groups:

A: Control Group

B: Massage Group, 15 minutes twice a day;

C: Massage and physical exercise group 15 minutes each, twice a day.

ELIGIBILITY:
Inclusion Criteria:

* low birth weight, less than 1500 grams
* weight of at least 1000 grams at time of entry into study
* must be at least one week of age
* must have relative medical stability
* gestational age between 28-32 weeks

Exclusion Criteria:

* infants with major congenital anomaly
* those that require mechanical ventilatory support
* those that are restricted in their movement or ability to undergo the intervention

Ages: 28 Weeks to 32 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2003-02; Primary Completion 2007-04 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Average daily weight gain. Length of hospital stay | From birth until time of hospital discharge

SECONDARY OUTCOMES:
Effect on heart rate and respirations | Birth until time of hospital discharge

CONTACTS AND LOCATIONS:
Overall Officials: Hany Z Aly, MD, Principal Investigator — George Washington University
Locations (1):
- George Washington University Hospital, Washington D.C., District of Columbia, United States